CLINICAL TRIAL: NCT03340363
Title: "Make It Fresh, For Less" Supermarket Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Duke University (Other); University of New England (Other); Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Eric B. Rimm, Professor of Epidemiology and Nutrition, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: BECR-111191
Record Dates: First submitted 2017-02-08; First posted 2017-11-13 (Actual); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Food Habits; Consumer Behavior
MeSH Terms: conditions — Feeding Behavior; Consumer Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- environmental change (Experimental): Shoppers were exposed to modifications to the supermarket environment to encourage selection of low-cost, kid-friendly meals
  Interventions: Behavioral: environmental change
- environmental change and messaging (Experimental): Shoppers were exposed to modifications to the supermarket environment and weekly messages via text or email to encourage selection of low-cost, kid-friendly meals
  Interventions: Behavioral: environmental change; Behavioral: messaging

INTERVENTIONS:
Behavioral: environmental change — 1. Offer kid-friendly, low-cost recipes in a prominent, high-traffic location.
  2. Offer healthy default ingredients (bundled ingredients promoted with recipes).
  3. Promote recipe ingredients with prominently displayed signage and images.
  4. Promote recipes in multiple locations throughout the store.
  Other Names: choice architecture; promotional campaign
Behavioral: messaging — Short, behavioral messages sent to participants via text message or email each week to promote the in-store environmental changes
  Arms: environmental change and messaging

SUMMARY:
The purpose of this study is to examine the impact of environmental modifications (choice architecture and a marketing campaign) in combination with weekly text messages on purchases of foods made by parents shopping in a large supermarket.

DETAILED DESCRIPTION:
The "Make It Fresh, For Less" Supermarket Pilot Study is a supermarket-based intervention developed by the Harvard T.H. Chan School of Public Health in collaboration with the nonprofit organization ChopChop Magazine (chopchopmagazine.org) and a large Northeastern supermarket chain. A promotional campaign advertising low-cost, kid-friendly meals was piloted in one store selected by the supermarket partner, with promotions rotating every 4 weeks during a 16-week intervention period. Parent shoppers were recruited (n=401) at the store and given a study loyalty card to track their transactions. At the start of the intervention, half of the participants were additionally randomized to receive weekly behavioral messages via text message or email. Supermarket purchases were assessed at baseline, during the 16-week intervention, and up to 6-weeks post-intervention.

Primary Aim 1: to examine the impact of a choice architecture intervention in combination with a promotional campaign on food purchases of parents shopping in a large supermarket. It is hypothesized that there will be an increase in selection of foods targeted by the promotional campaign when physical modifications are made.

Primary Aim 2: to examine the impact of weekly behavioral messages in combination with an environmental change intervention on food purchases of parents shopping in a large supermarket. It is hypothesized that there will be a greater increase in selection of foods targeted by the promotional campaign among participants receiving the messages compared to participants exposed to the environmental change intervention alone.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* English-speaking
* Live with a child 18 years of age or younger
* Do more than 50% of shopping at the study store
* Primary shopper in the household

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 401 (Actual)
Dates: Start 2015-10-08 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
Change in weekly purchases of recipe components (Selection of items bundled with each recipe) during four, 4-week promotional campaigns | Baseline, during intervention (4 weeks each) and up to 6 weeks post-intervention
  Purchase of recipe ingredients

SECONDARY OUTCOMES:
Change in weekly purchases of other food categories (substitution of recipe ingredients for other foods) | Baseline, during intervention (4 weeks each) and up to 6 weeks post-intervention
  Substitution of recipe ingredients for other foods
Differential change in weekly purchases of recipe components by SNAP-eligibility | Baseline, during intervention (4 weeks each) and up to 6 weeks post-intervention
  Stratification by SNAP-eligibility, recipe components
Differential change in weekly purchases of other food groups (substitution) by SNAP-eligibility | Baseline, during intervention (4 weeks each) and up to 6 weeks post-intervention
  Stratification by SNAP-eligibility, other food groups
Acceptability of intervention (self-reported survey measures) | Up to 6 weeks post-intervention
  Shopper responses to survey questions asking participants to rate the acceptability of each recipe (taste, cost, difficulty, perceptions of children's preferences) on a Likert scale from 1-5.
Recall of intervention (self-reported survey measures) | Up to 6 weeks post-intervention
  Shopper responses to survey questions regarding aided and unaided recall. Unaided recall asks shoppers to choose the best description of what they saw in the store and aided recall asks shoppers whether they remember seeing various elements of the display in the store (yes, no, not sure). These measures will be combined to report the proportion of shoppers who recalled each component of the intervention either through aided or unaided means.
Adoption of intervention (self-reported survey measures) | Up to 6 weeks post-intervention
  Shopper responses to survey questions asking whether the shopper made each recipe in the display.
Reach of intervention (direct observation measures) | During intervention (4 weeks each)
  Observation of shopper interactions with promotional campaign (count of number of shoppers who passed the display, looked at the display, and took an item from the display).
Fidelity to intended intervention (direct observation measures) | During intervention (4 weeks each)
  Monthly random site visits to assess presence or absence of each element of the display (placards, poster, recipe cards, intended ingredients, store banners).

IPD SHARING:
Plan to Share IPD: No